CLINICAL TRIAL: NCT01948297
Title: A Phase I, Gene Alteration-based, Open Label, Multicenter Study of Oral Debio 1347 (CH5183284) in Patients With Advanced Solid Malignancies, Whose Tumours Have an Alteration of the FGFR 1, 2 or 3 Genes
Brief Title: Debio 1347-101 Phase I Trial in Advanced Solid Tumours With Fibroblast Growth Factor Receptor (FGFR) Alterations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debio 1347-101; 2013-000316-19 (EudraCT Number)
Record Dates: First submitted 2013-08-26; First posted 2013-09-23 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumours
MeSH Terms: interventions — CH5183284

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Adaptive doses of Debio1347 (CH5183284) - (10 mg to 210 mg/day) until the recommended dose (RD) is determined.
  Interventions: Drug: Debio1347 (CH5183284)
- Part B (Experimental): Participants with various tumours receive Debio1347 (CH5183284) orally at the recommended dose established during Part A.
  Interventions: Drug: Debio1347 (CH5183284)

INTERVENTIONS:
Drug: Debio1347 (CH5183284) — Debio1347 (CH5183284) tablets for oral administration
  Other Names: CH5183284

SUMMARY:
This study is primarily designed to assess the safety and the tolerability of Debio1347 (CH5183284) in patients with advanced solid malignancies, whose tumours have an alteration of the Fibroblast Growth Factor Receptor (FGFR) 1, 2 or 3 genes, for whom standard treatment does not exist or is not indicated.

The main objective of Part A is to identify the dose-limiting toxicities (DLTs) and estimate the maximum tolerated dose (MTD) based on the safety and tolerability of Debio1347 orally administered daily to these patients, in order to determine the recommended dose.

The main objective of Part B is to evaluate the safety profile at the recommended dose, in a larger cohort of these patients.

ELIGIBILITY:
Inclusion Criteria

* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related to food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding)
  3. the analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-08; Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Part A: Percentage of Participants With Dose-Limiting Toxicities (DLTs) From Debio 1347 | within approximately 18 months
Part B: Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs) | within 2 years of starting treatment
Part B: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | within 2 years of starting treatment
Part B: Severity of Treatment-Emergent AEs | within 2 years of starting treatment
  Categories: NCI-Common Terminology Criteria for Adverse Events (CTCAE) version 4 severity criteria
Part B: Severity of Laboratory Abnormalities | within 2 years of starting treatment
  Categories: NCI-Common Terminology Criteria for Adverse Events (CTCAE) version 4 severity criteria

SECONDARY OUTCOMES:
Part A: Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs) | within 2 years of starting treatment
Part A: Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | within 2 years of starting treatment
Part A: Severity of Treatment-Emergent AEs | within 2 years of starting treatment
  Categories: NCI-CTCAE version 4 severity criteria
Part A: Severity of Laboratory Abnormalities | within 2 years of starting treatment
  Categories: NCI-CTCAE version 4 severity criteria
Part A and Part B: Percentage of Participants With Treatment Discontinuations or Modifications due to AEs and Laboratory Abnormalities | within 2 years of starting treatment
Part A and Part B: Number of Participants With Change From Baseline in Blood Pressure (BP) | within 2 years of starting treatment
  Change in BP will be evaluation based on three criteria- "Change to Low" (decrease from pre-treatment > 20 millimeter of mercury [mmHg]), "No change" (change from pre-treatment within ± 20 mmHg) and "Change to High" (increase from pre-treatment > 20 mmHg).
Part A and Part B: Number of Participants With Change From Baseline in Pulse Rate | within 2 years of starting treatment
  Number of participants with change of more than 20 beats per minute from baseline will be reported.
Part A and Part B: Number of Participants With Change From Baseline in Electrocardiogram (ECG) Parameters | within 2 years of starting treatment
  ECG parameters will include PR, RR, QRS, QTcB and QTcF intervals.
Part A and Part B: Change From Baseline in Left Ventricular Ejection Fraction (LVEF) | within 2 years of starting treatment
Part A and Part B: Change From Baseline in Eastern Cooperative Oncology Group Performance Status (ECOG PS) | within 2 years of starting treatment
Part A: Number of Participants With Tumour Response, According to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 Criteria | within 2 years of starting treatment
  Includes: Best overall response, disease control, tumour size
Part B: Number of Participants With Tumour Response, According to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 Citeria or Response Assessment in Neuro-Oncology (RANO) (for glioblastoma participants) | within 2 years of starting treatment
  Includes: Best overall response, disease control, tumour size
Part A and Part B: Progression-Free Survival Rate After Treatment Initiation | within 2 years of starting treatment
  Categories: overall, 6 months, 1 year, 2 years
Part A and Part B: Number of Participants With Changes in Ophthalmological Exams | within 2 years of starting treatment
  Opthalmological exams includes visual acuity testing, slit-lamp ophthalmoscopy and indirect ophthalmoscopy.
Part A: Area Under Concentration-Time Curve (AUC) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Concentration at the end of a Dosing Interval (Ctrough) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Maximum Observed Concentration (Cmax) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Time of Maximum Concentration (tmax) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Apparent Terminal Half-Life (t1/2) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Mean Residence Time (MRT) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Apparent Clearance (CL/F) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Apparent Volume of Distribution (Vz/F) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Accumulation Ratios (RAC) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Linearity Index (LI) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part A: Peak-to-Trough fluctuation (PTF) Following Single- and Repeated-Dose Administration of Debio 1347 | Day -9, Day -2, Day 28; Ctrough on Day 8, Day 15, Day 22 of Cycle 1, and on Day 1 of Cycle 2 and Cycle 3
Part B: Area Under Concentration-Time Curve (AUC), Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Concentration at the end of a Dosing Interval (Ctrough) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Maximum Observed Concentration (Cmax) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Time of Maximum Concentration (tmax) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Apparent Terminal Half-Life (t1/2) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Mean Residence Time (MRT) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Apparent clearance (CL/F) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Apparent Volume of Distribution (Vz/F) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Peak-to-Trough Fluctuation (PTF) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Renal Clearance (CLR) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Percentage of the Dose Excreted in Urine (Ae%) Following Repeated-Dose Administration of Debio 1347 in the PK Subset | Day 28
Part B: Ctrough in all Participants | Day 8, Day 15, Day 22 of Cycle 1, and Day 1 of Cycle 2 and Cycle 3

CONTACTS AND LOCATIONS:
Locations (8):
- United States (4):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan-Kettering Hospital, New York, New York
  - The University of Texas; MD Anderson Cancer Center, Houston, Texas
- National Cancer Center Singapore, Singapore, Singapore
- Seoul National University Hospital, Seoul, South Korea
- Vall d'Hebron University Hospital, Barcelona, Spain
- Taipei Medical University Hospital, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.debiopharm.com